CLINICAL TRIAL: NCT02189954
Title: Effect of Laryngeal Mask Cuff Pressure on Postoperative Pharyngolaryngeal Complications in Geriatric Patients
Brief Title: Effect of Laryngeal Mask Cuff Pressure in Geriatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 269-GOA
Record Dates: First submitted 2014-06-28; First posted 2014-07-15 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Anaesthesia
Keywords: elderly; laryngeal masks; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Routine Care (Active Comparator): The placement according to the manufacturer's instructions.
  Interventions: Procedure: The placement according to the manufacturer's instructions
- Group Pressure Limiting (Experimental): Cuff inner pressure was held below 44 mmHg
  Interventions: Procedure: Cuff inner pressure was held below 44 mmHg

INTERVENTIONS:
Procedure: The placement according to the manufacturer's instructions — Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique®(LMU)) was lubricated with a water-based gel and the cuff was completely deflated. After induction when BIS values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than five years experience
  Arms: Group Routine Care
Procedure: Cuff inner pressure was held below 44 mmHg — cuff pressure limitation (Group Pressure Limiting (PL), n=45) cuff inner pressure was held below 60 cmH2O (44 mmHg)
  Arms: Group Pressure Limiting

SUMMARY:
Laryngeal Mask is widely used for air-way management during anaesthesia. Pharyngolaryngeal morbidity linked to laryngeal mask use is related to correct choice of mask size, placement technique, placement of the laryngeal mask in the correct position on the larynx, cuff volume and cuff pressure. It has been stated that keeping laryngeal mask cuff pressure below 45 mmHg (60 centimeter of water(cmH2O) ) can prevent pharyngolaryngeal morbidity related to laryngeal mask (throat pain, dysphonia, dysphagia) and shown that using a manometer after Laryngeal Mask Unique placement to limit pressure within the cuff can reduce this morbidity by nearly 70%. Studies commenting on pharyngolaryngeal morbidity generally do not choose a certain age group and cover stages including very young and middle-aged groups. In the literature only one similar study on the geriatric age group was found.

The aim of this study is to compare the postoperative pharyngolaryngeal morbidity in a group with cuff pressure held to 44 mmHg (60 cmH2O with a manometer and a group with Laryngeal Mask cuff inflated without reference to pressure in the geriatric age group with indications for Laryngeal Mask Unique placement.

DETAILED DESCRIPTION:
This study received permission from Dokuz Eylül University Medical Faculty Non-Interventional Ethics Committee and informed consent was obtained from the patients. Ninety patients above the age of 65 with American Society of Anesthesiologists (ASA) physiological classification group I-III, undergoing elective surgery and with indications for laryngeal mask placement participated in this prospective, randomized and double blind study.

Patients taken to the operating room were given standard monitoring (ECG, pulse oxymetry, non-invasive blood pressure) and BIS monitoring [BIS-Vista ™ (Aspect Medical Systems, USA)] before anesthesia induction.

After patients were preoxygenated with 6 L/min oxygen through a face mask for 3 minutes anesthesia induction was provided by 0.02 mg/kg midazolam, 1-2 µg/kg fentanyl and 1-2 mg/kg propofol. During respiration Airway was not used, unless there was ventilation difficulty with the face mask. Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique® (LMU)) was lubricated with a water-based gel and the cuff was completely deflated. After induction when bispectral index (BIS) values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than five years experience. The placement method was according to the manufacturer's instructions. All patients were respirated by a breathing circuit with heat and moisture filter.

After the laryngeal mask was inserted the cases were manually respirated so peak inspiratory pressure was less than 20 cmH2O and the cuff of both groups was inflated with a 20 ml injector until the leak sound ceased. To evaluate ventilation the capnogram showed square wave forms and the patients' chest movements were observed, in unsuccessful situations the procedure was repeated. During attempts depending on the patients' reactions and with the requirement of keeping BIS values between 40 and 60, an additional dose of 0.5 mg/kg propofol was administered.

After Laryngeal Mask was determined and when anesthetic depth was sufficient (BIS 40-60) the inner pressure of the LMU cuff was measured and recorded by a manometer (cuff pressure manometer, Rusch, Germany). Later groups were divided in two using a random number table. In the group with cuff pressure limitation (Group Pressure Limiting (PL), n=45) cuff inner pressure was held below 60 cmH2O (44 mmHg), while the routine group (Group Routine Care, n=45) pressure was only recorded.

Anesthesia was maintained by 50% O2:50% air mix with 1.5-2.5% sevoflurane, with sevoflurane concentration and additional fentanyl doses arranged to keep BIS between 40 and 60. All patients were respirated with positive pressure ventilation tidal volume 7-8 ml/kg, inspiring: expiring rate 1:2, respiration frequency on the capnograph end tidal carbon dioxide held between 30-35 mmHg. Oropharyngeal leak pressure measurement was recorded as the pressure value when a leak sound was heard from the mouth after the expiring valve was closed and fresh gas flow was reduced to 3 L/min. Immediately after the laryngeal mask was inserted, every 5 minutes in the first half hour and every 15 minutes after that, tidal volume, mean airway pressure, end tidal carbon dioxide levels and peripheral oxygen saturation values were recorded. If the operation lasted more than one hour a second manometric measurement was taken and stable values were maintained.

After the operation, the LMU's were removed when the patients were awake and could open their mouths on an oral command and unless necessary, aspiration was not applied.After anesthesia the patients were monitored in the recovery unit and analgesia was provided by 5-10 mg intravenous dolantin titration. A researcher blind to the groups recorded throat pain, voice loss and difficulty swallowing in the 1st and 24th hour, classifying as Likert scale ranges from 1 (none) to 4 (severe). Cases developing rare complications of recurrent laryngeal nerve, hypoglossal nerve and lingual nerve paralysis were recorded. The cases were brought to the ward when Aldrete scoring criteria were appropriate. Cases discharged early from the ward had 24th hour evaluation by telephone communication.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 65
* ASA I-III
* Undergoing elective surgery

Exclusion Criteria:

* Patients with recent history of upper respiratory infection
* Obese patients with body-mass index above 35 kg/m2
* Symptomatic hiatus hernia
* Severe gastroesophageal reflux
* Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FERİM GÜNENÇ, M.D., Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmi̇r, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Routine Care: The placement according to the manufacturer's instructions.
  The placement according to the manufacturer's instructions: Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique® (LMU) was lubricated with a water-based gel and the cuff was completely deflated. After induction when bispectral index (BIS) values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than five years experience
- Group Pressure Limiting: Cuff inner pressure was held below 44 mmHg
  Cuff inner pressure was held below 44 mmHg: cuff pressure limitation (Group Pressure Limiting (PL)), n=45) cuff inner pressure was held below 60 centimeter of water (cmH2O) (44 mmHg)
Period: Overall Study
Arm/Group | Group Routine Care | Group Pressure Limiting
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group Routine Care: The placement according to the manufacturer's instructions.
  The placement according to the manufacturer's instructions: Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique®) was lubricated with a water-based gel and the cuff was completely deflated. After induction when BIS values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than five years experience
- Group Pressure Limiting: Cuff inner pressure was held below 44 mmHg
  Cuff inner pressure was held below 44 mmHg: cuff pressure limitation (Group PL, n=45) cuff inner pressure was held below 60 cmH2O (44 mmHg)
- Total: Total of all reporting groups
Arm/Group | Group Routine Care | Group Pressure Limiting | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (5.4) | 72.8 (6.2) | 72.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  Turkey | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pharyngolaryngeal Morbidity Postoperative 1.Hour
Description: The primary outcome was a composite endpoint of any pharyngolaryngeal complications such as sore throat, dysphonia and dysphagia according to Likert scale ranges from 1 (none) to 4 (severe) at postoperative 1.hour
Time Frame: Postoperative 1.hour
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group Routine Care | Group Pressure Limiting
Number analyzed (Participants) | 45 | 45
units on a scale | 1 [1 to 4] | 1 [1 to 2]

2. Secondary Outcome: Postoperative Pharyngolaryngeal Morbidity at Postoperative 24.Hour
Description: The primer outcome was a composite endpoint of any pharyngolaryngeal complications such as sore throat, dysphonia and dysphagia according to Likert scale ranges from 1 (none) to 4 (severe) at postoperative 24.hour
Time Frame: Postoperative 24.hour
Population: Chi Square Test for categorical variables, for constant variables t test when suitable for normal distribution and when unsuitable for normal distrubition Mann Whitney U have been used for analysis. p < 0.05 was considered significant.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group Routine Care | Group Pressure Limiting
Number analyzed (Participants) | 45 | 45
units on a scale | 1 [1 to 3] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Group Routine Care vs Group Pressure Limiting; Test type: Superiority or Other; p < 0.05, Chi-squared
Statistical Analysis 2: Comparison: Group Routine Care vs Group Pressure Limiting; Test type: Superiority or Other; p < 0.05, Mann Whitney U

ADVERSE EVENTS:
Arm/Group | Group Routine Care | Group Pressure Limiting
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
Limitations of our study include the lack of imaging with a fiberoptic bronchoscope after LMU placement and not evaluating the position in the hypopharynx of the supraglottic airway device in the geriatric age group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No